CLINICAL TRIAL: NCT07082530
Title: Labor Induction in Low-risk Women at 39 Weeks of Gestation to Reduce Cesarean Rate: A Pilot Randomized Trial in China
Brief Title: A Pilot Study of Induction at 39 Weeks to Reduce Cesarean in Low - Risk Women in China
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-20250211-R
Record Dates: First submitted 2025-06-25; First posted 2025-07-24 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Cesarean Delivery
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induction group (Experimental): Labor induction at 39 weeks 0 days to 39 weeks 4 days
  Interventions: Procedure: Labor Induction at 39 Weeks
- Control group (Active Comparator): Expectant management until spontaneous labor or induction at 41 weeks
  Interventions: Procedure: Expectant management

INTERVENTIONS:
Procedure: Labor Induction at 39 Weeks — Labor induction at 39 weeks 0 days to 39 weeks 4 days
  Arms: Induction group
Procedure: Expectant management — Expectant management until spontaneous labor or induction at 41 weeks.
  Arms: Control group

SUMMARY:
The investigators are committed to identifying the optimal timing of delivery for low-risk pregnancies. While current guidelines typically recommend induction at 41 weeks, emerging evidence suggests that elective induction at 39 weeks may lead to improved maternal and neonatal outcomes. The U.S.-based ARRIVE trial demonstrated that induction at 39 weeks significantly reduced cesarean delivery rates compared to expectant management, and a similar randomized controlled trial (French-ARRIVE) is ongoing in France. However, population-specific evidence for the Chinese population remains lacking.

This study is designed to establish a prospective cohort of low-risk pregnant women in China, comparing the effects of induction at 39 weeks, induction at 41 weeks, and expectant management on cesarean section rates and other maternal and neonatal outcomes. In addition, multi-omics technologies will be employed to analyze cord blood samples-including metabolomics and proteomics-to identify early biomarkers potentially associated with long-term child health. The study will begin with a pilot phase to assess feasibility and inform operational strategies for large-scale implementation.

The ultimate goal of this project is to generate evidence tailored to the Chinese population to support more individualized decision-making, improve clinical outcomes, and enhance maternal and neonatal safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Singleton pregnancy or twin pregnancy reduced to singleton before 14 weeks.
3. Gestational age of 38 weeks 6 days or 39 weeks 0 days at randomization.
4. Eligible for vaginal delivery with a desire for vaginal birth.
5. Reliable gestational age determination.
6. Maternal and fetal conditions assessed as favorable by at least two senior obstetricians, with no indications requiring delivery before 41 weeks.
7. Ability to understand study information and provide informed consent.

Exclusion Criteria:

1. First ultrasound estimate >13 weeks 6 days.
2. Planned induction before 41 weeks.
3. Planned cesarean delivery or contraindications to vaginal delivery.
4. Already delivered, in labor, or ruptured membranes at enrollment.
5. Placenta previa, vasa previa, placenta accreta, or placental abruption.
6. Contraindications to induction (e.g., cervical cancer, history of uterine rupture, genital tract malformations, abnormal fetal position, cord prolapse).
7. Active vaginal bleeding exceeding spotting.
8. History of cesarean delivery or uterine/cervical surgery.
9. Cervical cerclage during this pregnancy.
10. Maternal conditions not suitable for expectant management beyond 39 weeks (e.g., pregestational diabetes, gestational diabetes requiring insulin, hypertensive disorders, intrahepatic cholestasis of pregnancy).
11. Fetal conditions not suitable for expectant management beyond 39 weeks (e.g., fetal death, major anomalies, growth restriction, macrosomia, anemia, oligohydramnios, polyhydramnios).
12. Maternal infections or positive screenings for sexually transmitted pathogens or group B Streptococcus.
13. Planned delivery at a non-study facility.
14. Participation in another intervention study affecting delivery management.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1074 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of cesarean section | Delivery day
  The proportion of deliveries completed by cesarean section

SECONDARY OUTCOMES:
Composite incidence of severe neonatal morbidity and perinatal mortality | Hospital discharge (Day 2-3)
  The composite incidence of any of the following:
  1. Antepartum, intrapartum, or neonatal death
  2. Intubation, continuous positive airway pressure (CPAP) or high-flow nasal cannula (HFNC) for ventilation or cardiorespiratory support within first 72 hours
  3. Apgar ≤ 3 at 5 minutes
  4. Neonatal encephalopathy
  5. Seizures
  6. Sepsis (presence of a clinically ill infant in whom systemic infection is suspected with a positive blood, cerebral spinal fluid (CSF), or catheterized/suprapubic urine culture; or, in the absence of positive cultures, clinical evidence of cardiovascular collapse or an unequivocal X-ray confirming infection).
  7. Pneumonia confirmed by X-ray or positive blood culture.
  8. Meconium aspiration syndrome
  9. Birth trauma (bone fractures, brachial plexus palsy, other neurologic injury, retinal hemorrhage, facial nerve injury)
  10. Intracranial hemorrhage or subgaleal hemorrhage
  11. Hypotension requiring pressor support
Emergency Cesarean Rate | Delivery day
  Cesarean delivery performed immediately or shortly after clinical decision due to imminent threat to the life of the mother or fetus
Category 1 Emergency Cesarean Rate | Delivery day
  Cesarean performed within approximately 30 minutes due to immediate life-threatening conditions (e.g., uterine rupture, severe fetal distress)
Category 2 Emergency Cesarean Rate | Delivery day
  Cesarean performed within 60-75 minutes due to urgent but not immediately life-threatening indications (e.g., progressive fetal distress, labor arrest)
Elective Cesarean Rate | Delivery day
  Planned cesarean performed at or after 39 weeks in the absence of emergency conditions, meeting all of the following:
  1. Surgery scheduled ≥24 hours before onset of labor;
  2. No spontaneous contractions or rupture of membranes;
  3. Clear medical indications (e.g., placenta previa, breech presentation) or maternal request.
Operative Vaginal Delivery | Delivery day
  The rate of vaginal deliveries assisted with instruments such as forceps or vacuum.
Gestational Age at Delivery | Delivery day
  Expressed in weeks and decimal days (e.g., 39 weeks + 5 days = 39.7 weeks)
Chorioamnionitis | Delivery day
  Incidence of chorioamnionitis, defined as a clinical diagnosis before delivery as: maternal body temperature rises (>38°C) with 1 or more of the following symptoms:
  1. Maternal tachycardia (>100 beats/min);
  2. Fetal tachycardia (>160 beats/min)
  3. Uterine tenderness and irritability
  4. Purulent or malodorous amniotic fluid or vaginal discharge
  5. Maternal leukocytosis (white blood cell count > 15000/mm3)
Third-or fourth-degree perineal laceration | Delivery day
  The incidence of third-or fourth-degree perineal laceration
Time from Randomization to Delivery | Delivery day
  Measured in hours
Postpartum hemorrhage | Hospital discharge (Day 2-3)
  Refer to the ARRIVE cohort, defined as any of the following situations:
  1. Transfusion
  2. Non-elective hysterectomy
  3. Use of two or more uterotonics other than oxytocin
  4. Other surgical interventions such as uterine compression sutures, uterine artery ligation, embolization and hypogastric ligation, balloon tamponade
  5. Curettage
Postpartum infection | Hospital discharge (Day 2-3)
  Refer to the ARRIVE cohort, defined as any of the following situations:
  1. Clinical diagnosis of endometritis
  2. Wound reopened for hematoma, seroma, infection or other reasons
  3. Cellulitis requiring antibiotics
  4. Pneumonia
  5. Pyelonephritis
  6. Bacteremia unknown source
  7. Septic pelvic thrombosis
ICU admission | Hospital discharge (Day 2-3)
  The proportion of admission to the ICU
Maternal death | Hospital discharge (Day 2-3)
  The incidence of maternal death
Preeclampsia/gestational hypertension | Hospital discharge (Day 2-3)
  The incidence of preeclampsia or gestational hypertension diagnosed during labor
Maternal venous thromboembolism | Hospital discharge (Day 2-3)
  Deep vein thrombosis or pulmonary embolism
Maternal pain | Hospital discharge (Day 2-3)
  Median patient-reported pain outcomes with a 10-point Likert scale
Birth weight | Delivery day
  The mean birth weight
Female gender | Delivery day
  The proportion of female offspring in terms of physiological gender
Macrosomia | Delivery day
  Birth weight > 4000g
Incidence of large for gestational age | Delivery day
  According to the infant's gender and gestational age, the birth weight exceeds the 90th percentile of infants of the same gestational age
Incidence of small for gestational age | Delivery day
  According to the infant's gender and gestational age, the birth weight is less than the 10th percentile of infants of the same gestational age
Apgar scores at 5 min | Delivery day
  Apgar score at 5 minutes after birth
Neonatal acidosis | Delivery day
  The incidence of neonatal acidosis defined as umbilical artery blood pH < 7.00
Shoulder dystocia | Delivery day
  The incidence of shoulder dystocia
Hyperbilirubinemia | Hospital discharge (Day 2-3)
  The incidence of hyperbilirubinemia requiring phototherapy or exchange transfusion
Transfusion of blood products or blood | Hospital discharge (Day 2-3)
  The incidence of neonatal transfusion of blood products or blood
Hypoglycemia incidence | Hospital discharge (Day 2-3)
  The incidence of hypoglycemia (blood glucose < 35mg/L) requiring intravenous treatment
Neonatal intensive care unit (NICU) admission | Hospital discharge (Day 2-3)
  The incidence of admission to the NICU
Physical measurement indicators | 42 days and 6 months
  Infant weight, length, head circumference, chest circumference, sitting height, upper arm circumference, subcutaneous fat, height-chest circumference index, crown-rump length/length
Growth balance indicators | 42 days and 6 months
  Weight-for-length, length-for-age, weight-for-age z scores of infants, calculated using the World Health Organization (WHO) tool, WHO Anthro Survey Analyser
Growth retardation | 42 days and 6 months
  Height standard deviation for age < mean-2S or percentile method < P3
Abnormal neurological examination | 42 days and 6 months
  The proportion of abnormal results in neurological examinations (hearing development, nerve reflexes)
Scores of Bayley Scales of Infant and Toddler Development | 42 days and 6 months
  Total score, cognitive scale score, language scale score, motor scale score, social-emotional scale score, adaptive behavior scale score
Scores of Ages & Stages Questionnaires®, Third Edition (ASQ-3) | 42 days and 6 months
  Total score, communication domain score, gross motor domain score, fine motor domain score, problem-solving domain score, personal-social domain score
Gut microbiota development | Meconium, first 48 hours, 7 days, 6 weeks and 6 months
  Microbiota richness, dominant species, species transferred from mother to child, sub-group functional trajectory changes of the dominant species in offspring, and the transmissibility of species number and function
Fecal metabolomic characteristics | Meconium, first 48 hours, 7 days, 6 weeks and 6 months
  Non-targeted metabolomic macroscopic differences, core metabolomic differences (including tryptophan, fatty acids), and differences in gut microbiota metabolites
Cord blood metabolomic characteristics | Delivery day
  Assessment of non-targeted metabolomic macroscopic differences and core metabolomic differences (including tryptophan, fatty acids) in cord blood plasma
Cord blood proteomic characteristics | Delivery day
  Analysis of the proteomic characteristics of cord blood whole blood to trace back the health status during the fetal period
Time from randomization to delivery | Delivery day
  Median time from randomization to birth of the fetus, measured in hours
Use of epidural analgesia | Delivery day
  Rate of epidural analgesia use
Time spent in the delivery room | Delivery day
  Median time spent in the delivery room, measured in hours
Length of postpartum hospital stay | Hospital discharge (Day 2-3)
  Median postpartum length of stay, measured in hours
Neonatal length of hospital stays | Hospital discharge (Day 2-3)
  Median neonatal hospital stays, measured in hours
Pre-insurance hospitalization cost | Hospital discharge (Day 2-3)
  Total hospitalization cost during delivery, before insurance reimbursement
Out-of-pocket hospitalization cost | Hospital discharge (Day 2-3)
  Out-of-pocket cost incurred during delivery hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Dan Zhang, Ph. D., Principal Investigator — Key Laboratory of Reproductive Genetics, Women's Hospital, Zhejiang University School of Medicine
Locations (1):
- Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang, China

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT07082530/Prot_SAP_002.pdf
  • Informed Consent Form (2025-06-04): https://cdn.clinicaltrials.gov/large-docs/30/NCT07082530/ICF_003.pdf